CLINICAL TRIAL: NCT03728764
Title: Growth and Safety of a Two-stage Feeding System in Preterm Infants: a Prospective, Non-randomized, Open-label, Single-arm Study
Brief Title: Growth and Safety of a Two-stage Feeding System in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17.14.INF
Record Dates: First submitted 2018-08-02; First posted 2018-11-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other)
  Interventions: Other: Preterm infant formula

INTERVENTIONS:
Other: Preterm infant formula — Preterm infants will receive Stage 1 investigative product as soon as possible after birth until when 1.8 kg of body weight is achieved. Preterm infants will receive stage 2 preterm formula from when 1.8 kg of body weight is achieved until 1 month after hospital discharge.

SUMMARY:
This study evaluates the safety and suitability of the two-stage feeding system in preterm infants.

DETAILED DESCRIPTION:
This open-label trial will be conducted in up to 74 preterm infants to evaluate the formula as it would typically be used in the neonatal care unit and to document the safety and suitability of the two-stage feeding system in terms of growth in comparison to recommended growth goals, feeding tolerance, biochemical parameters, and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from the parents/legally acceptable representative (LAR).
2. Infant's birth weight ≤1500 g and appropriate for gestational age (AGA) as defined by weight ≥10 percentile and ≤90 percentile on the Fenton growth chart.
3. Infant's gestational age ≥ 27 weeks and ≤ 32 weeks.
4. Infant is clinically stable.
5. Infants are eligible to start experimental formula within the first 5 days (≤120 hours) of life.

Exclusion Criteria:

1. Parents not willing / not able to comply with the requirements of study protocol.
2. Infants experiencing early onset sepsis.
3. Major congenital or chromosomal abnormality known to affect growth.
4. Preterm infants experiencing liver failure.
5. Peri-/intra-ventricular haemorrhage.
6. Infant requiring prolonged (more than 3 doses) of steroid treatment.
7. Infants' participation in another interventional clinical trial.

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Growth of preterm infants | from FEF Day 1 to when infant reaches 1800 g (on average between 4 to 6 weeks after birth) or hospital discharge (on average 7 weeks after birth), whichever comes earlier
  Weight gain

SECONDARY OUTCOMES:
Other growth parameter at other time points | from Pre-FEF Day 1 to FEF Day 1, and then weekly from FEF Day 1 until hospital discharge (on average 7 weeks after birth) and at 30-days PD.
  Changes in weight gain (in g/day)
Other growth parameter | from Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth) and at 30-days PD.
  Changes in length (cm)
Other growth parameter | from Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth) and at 30-days PD.
  Head circumference (HC) (cm)
Other growth parameter | from Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth) and at 30-days PD ..
  Corresponding z-scores and changes in z-scores expressed using Fenton growth chart will be analyzed
Feeding intake: | daily between Pre-FEF day 1 and hospital discharge (on average 7 weeks after birth)
  Neonatal unit feeding questionnaire capturing milk intake (Volume in ml/range from 0 to 1000ml)
Feeding tolerance: | weekly between FEF Day 1 and hospital discharge (on average 7 weeks after birth)
  Tolerance to feeding regimen through neonatal unit questionnaire. Questionnaire assessing stool consistency (watery, mushysoft, runny, formed, hard); stool frequency (range from 0-20 times a day); Bloody stool (yes or no).
Feeding intake: | Daily during 30 days after hospital discharge
  Parent-reported questionnaire capturing milk intake (Volume in ml/range from 0 to 1000ml)
Feeding tolerance: | during the three days prior to the 30-day PD visit
  Tolerance to feeding through parent-reported questionnaire. Questionnaire assessing stool consistency (watery, mushysoft, runny, formed, hard); stool frequency (range from 0-20 times a day); Bloody stool (yes or no).
Neonatal unit routine blood collection for safety assessment (serum blood levels of blood urea nitrogen (BUN), creatinine, albumin, pre albumin) | will be obtained at Enrolment (baseline), if possible, Pre-FEF Day 1, FEF Day1, thereafter weekly until hospital discharge (on average 7 weeks after birth)., and lastly at 30 days post-discharge.
  Clinical abnormal values will be captured as part of adverse event reporting.
Number of AEs reported for safety assessment | from the time the mother has consented to the infant's participation in the study soon after birth but no later than 5 days of age after birth until the 30 days PD visit in the clinic.
  through investigator-confirmed AE reporting

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospital in Pilsen, Pilsen, Czechia
- Children's University Hospital, Krakow, Poland
- Slovakia (2):
  - University Hospital in Martin, Martin
  - Fakultná nemocnica s poliklinikou, Nové Zámky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwinta P, Lazarova S, Demova K, Chen Y, Hartweg M, Krattinger LF, Fumero C, Buczynska A, Durlak W, Uhrikova Z, Kozar M, Samuel TM, Zibolen M. Effects of two-stage preterm formulas on growth, nutritional biomarkers, and neurodevelopment in preterm infants. Front Pediatr. 2024 Nov 22;12:1427050. doi: 10.3389/fped.2024.1427050. eCollection 2024. PMID 39649400